CLINICAL TRIAL: NCT06099223
Title: Open-Label Randomized Controlled Trial to Assess Preoperative Acupuncture for Patients Undergoing Total Knee or Hip Arthroplasty
Brief Title: Preoperative Acupuncture for Total Knee or Hip Arthroplasty
Acronym: (Acupuncture)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Pranjali P Kainkaryam, MD, Principal Investigator, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HHC-2021-0348
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Knee Arthropathy; Hip Arthropathy; Anxiety
Keywords: Acupuncture; Total Knee Arthroplasty; Total hip arthroplasty; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, unblinded, randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Acupuncture (Experimental): Preoperative acupuncture
  Interventions: Device: Acupuncture needles
- Control (No Intervention): No acupuncture

INTERVENTIONS:
Device: Acupuncture needles — The acupuncture intervention includes a combination of auricular and body acupuncture. The auricular points used are Shen men, Zero point, Tranquilizer point, and Master cerebral.
  The body points used are the wrist PC6.
  Other Names: DBC™ Detox-5 Acupuncture Needles (SKU: DTX.20X13) and ure needles o 1) SEIRIN J-Type Acupuncture Needles (SKU: SJ.18X30)
  Arms: Acupuncture

SUMMARY:
Open-label, randomized controlled trial to determine the effect of preoperative acupuncture on preoperative anxiety and postoperative pain for high-anxiety patients undergoing total hip or knee arthroplasty. The hypothesis is that preoperative acupuncture will reduce preoperative anxiety, reduce postoperative pain, reduce postoperative nausea and vomiting, reduce opioid consumption, and improve patient satisfaction.

DETAILED DESCRIPTION:
Acupuncture has been extensively practiced and studied worldwide, particularly as a part of Eastern medicine, but it is a relatively uncommon therapy offered in Western medical institutions, such as those in the United States. Considering the commonly cited benefits of acupuncture, such as reduced anxiety and pain, hospitals throughout the United States have the opportunity to implement acupuncture as a cost-effective and safe technique for improving surgical outcomes.

Acupuncture administered in the preoperative period can be particularly effective for reducing preoperative anxiety, postoperative pain, postoperative opioid consumption, and postoperative nausea and vomiting. Consequently, preoperative acupuncture can improve patient satisfaction and decrease hospital costs. However, due to a lack of implementation and experience, further research is needed to establish the safety and efficacy of preoperative acupuncture in United States medical practices.

At the Bone-and-Joint Institute at Hartford Hospital, where this study is proposed, a quality study on total knee or hip arthroplasty patients found that 21% of its monthly patients were "high-anxiety" according to the Amsterdam Preoperative Anxiety and Information Scale (APAIS). Thus, there is a significant population of patients who would benefit from a procedure to reduce preoperative anxiety at our facility.

This proposal is for a prospective, open-label, randomized controlled trial to determine the effect of preoperative acupuncture on preoperative anxiety and postoperative pain for high-anxiety patients undergoing total hip or knee arthroplasty. The hypothesis is that preoperative acupuncture will reduce preoperative anxiety and postoperative pain as well as reduce postoperative nausea and vomiting and opioid consumption and improve patient satisfaction. The study population is to include adult patients undergoing lower extremity total joint arthroplasty, including hip and knee joints, at the Bone-and-Joint Institute at Hartford Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Female (age 52 to 85) or male (age 18-85) patients undergoing Total Knee Arthroplasty or Total Hip Arthroplasty at the Bone-and Joint Institute at Hartford Hospital
* Patients classified as high-anxiety based on having a score of >10 on the Amsterdam Preoperative Anxiety and Information Scale (APAIS-A-T). The APAIS-A-T is a modified survey that reliably quantifies total preoperative anxiety using summed scores for anesthesia and surgery-related anxiety; a minimum score of 11 is the most accurate cutoff to identify patients with anxiety

Exclusion Criteria:

* Unable to give consent
* Uncontrolled diabetes (HbA1c ≥ 8.0%)
* Infection at any of the acupuncture points
* Known allergy to metals
* Abnormal laboratory blood work values (INR>1.5, if available; platelet count <70,000, if available)
* Patients with active ongoing coagulopathy based on lab data (INR >1.5) and/or on current anticoagulant use which increases bleeding risk.
* Non-English speaking
* Revision TKA or THA
* Women of reproductive age or under the age of 52 years old, as acupuncture is not recommended during pregnancy. They were excluded due to the potential conflict between our institute's standard timing for pregnancy tests on the day of surgery and the scheduled preoperative acupuncture session for the study, to avoid unwanted delays in the operating room schedule.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women aged 52-85 were included. women under 52 were excluded due to the potential conflict between our institute's standard timing for pregnancy tests on the day of surgery and the scheduled preoperative acupuncture session for the study, to avoid unwanted delays in the operating room schedule.
Enrollment: 60 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bone and Joint Institute- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chernyak GV, Sessler DI. Perioperative acupuncture and related techniques. Anesthesiology. 2005 May;102(5):1031-49; quiz 1077-8. doi: 10.1097/00000542-200505000-00024. PMID 15851892
- [Background] Lu DP, Lu GP. An Historical Review and Perspective on the Impact of Acupuncture on U.S. Medicine and Society. Med Acupunct. 2013 Oct;25(5):311-316. doi: 10.1089/acu.2012.0921. PMID 24761180
- [Background] Crespin DJ, Griffin KH, Johnson JR, Miller C, Finch MD, Rivard RL, Anseth S, Dusek JA. Acupuncture provides short-term pain relief for patients in a total joint replacement program. Pain Med. 2015 Jun;16(6):1195-203. doi: 10.1111/pme.12685. Epub 2015 Jan 13. PMID 25586769
- [Background] Kotani N, Hashimoto H, Sato Y, Sessler DI, Yoshioka H, Kitayama M, Yasuda T, Matsuki A. Preoperative intradermal acupuncture reduces postoperative pain, nausea and vomiting, analgesic requirement, and sympathoadrenal responses. Anesthesiology. 2001 Aug;95(2):349-56. doi: 10.1097/00000542-200108000-00015. PMID 11506105
- [Background] Lao L, Bergman S, Hamilton GR, Langenberg P, Berman B. Evaluation of acupuncture for pain control after oral surgery: a placebo-controlled trial. Arch Otolaryngol Head Neck Surg. 1999 May;125(5):567-72. doi: 10.1001/archotol.125.5.567. PMID 10326816
- [Background] Mejuto-Vazquez MJ, Salom-Moreno J, Ortega-Santiago R, Truyols-Dominguez S, Fernandez-de-Las-Penas C. Short-term changes in neck pain, widespread pressure pain sensitivity, and cervical range of motion after the application of trigger point dry needling in patients with acute mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Apr;44(4):252-60. doi: 10.2519/jospt.2014.5108. Epub 2014 Feb 25. PMID 24568260
- [Background] Mikashima Y, Takagi T, Tomatsu T, Horikoshi M, Ikari K, Momohara S. Efficacy of acupuncture during post-acute phase of rehabilitation after total knee arthroplasty. J Tradit Chin Med. 2012 Dec;32(4):545-8. doi: 10.1016/s0254-6272(13)60068-0. PMID 23427386
- [Background] Tsang RC, Tsang PL, Ko CY, Kong BC, Lee WY, Yip HT. Effects of acupuncture and sham acupuncture in addition to physiotherapy in patients undergoing bilateral total knee arthroplasty--a randomized controlled trial. Clin Rehabil. 2007 Aug;21(8):719-28. doi: 10.1177/0269215507077362. PMID 17846072
- [Background] Usichenko TI, Dinse M, Hermsen M, Witstruck T, Pavlovic D, Lehmann C. Auricular acupuncture for pain relief after total hip arthroplasty - a randomized controlled study. Pain. 2005 Apr;114(3):320-327. doi: 10.1016/j.pain.2004.08.021. PMID 15777857
- [Background] Usichenko TI, Lehmann Ch, Ernst E. Auricular acupuncture for postoperative pain control: a systematic review of randomised clinical trials. Anaesthesia. 2008 Dec;63(12):1343-8. doi: 10.1111/j.1365-2044.2008.05632.x. PMID 19032304
- [Background] Zhang Y, Zhang L, Lu M. [Acupuncture combined with femoral nerve block for postoperative analgesia after total knee arthroplasty and functional rehabilitation: a randomized controlled trial]. Zhongguo Zhen Jiu. 2018 Mar 12;38(3):251-5. doi: 10.13703/j.0255-2930.2018.03.006. Chinese. PMID 29701041
- [Background] Lewis GN, Rice DA, McNair PJ, Kluger M. Predictors of persistent pain after total knee arthroplasty: a systematic review and meta-analysis. Br J Anaesth. 2015 Apr;114(4):551-61. doi: 10.1093/bja/aeu441. Epub 2014 Dec 26. PMID 25542191
- [Background] Bae H, Bae H, Min BI, Cho S. Efficacy of acupuncture in reducing preoperative anxiety: a meta-analysis. Evid Based Complement Alternat Med. 2014;2014:850367. doi: 10.1155/2014/850367. Epub 2014 Sep 2. PMID 25254059
- [Background] Usichenko TI, Dinse M, Lysenyuk VP, Wendt M, Pavlovic D, Lehmann C. Auricular acupuncture reduces intraoperative fentanyl requirement during hip arthroplasty--a randomized double-blinded study. Acupunct Electrother Res. 2006;31(3-4):213-21. doi: 10.3727/036012906815844265. PMID 17608061
- [Background] Wetzel B, Pavlovic D, Kuse R, Gibb A, Merk H, Lehmann C, Wendt M, Usichenko TI. The effect of auricular acupuncture on fentanyl requirement during hip arthroplasty: a randomized controlled trial. Clin J Pain. 2011 Mar-Apr;27(3):262-7. doi: 10.1097/AJP.0b013e3181fd516c. PMID 21346689
- [Background] Li M, Xing X, Yao L, Li X, He W, Wang M, Li H, Wang X, Xun Y, Yan P, Lu Z, Zhou B, Yang X, Yang K. Acupuncture for treatment of anxiety, an overview of systematic reviews. Complement Ther Med. 2019 Apr;43:247-252. doi: 10.1016/j.ctim.2019.02.013. Epub 2019 Feb 16. PMID 30935538
- [Background] Ali A, Lindstrand A, Sundberg M, Flivik G. Preoperative Anxiety and Depression Correlate With Dissatisfaction After Total Knee Arthroplasty: A Prospective Longitudinal Cohort Study of 186 Patients, With 4-Year Follow-Up. J Arthroplasty. 2017 Mar;32(3):767-770. doi: 10.1016/j.arth.2016.08.033. Epub 2016 Sep 3. PMID 27692782
- [Background] Ayers DC, Franklin PD, Ploutz-Snyder R, Boisvert CB. Total knee replacement outcome and coexisting physical and emotional illness. Clin Orthop Relat Res. 2005 Nov;440:157-61. doi: 10.1097/01.blo.0000185447.43622.93. PMID 16239800
- [Background] Bachmeier CJ, March LM, Cross MJ, Lapsley HM, Tribe KL, Courtenay BG, Brooks PM; Arthritis Cost and Outcome Project Group. A comparison of outcomes in osteoarthritis patients undergoing total hip and knee replacement surgery. Osteoarthritis Cartilage. 2001 Feb;9(2):137-46. doi: 10.1053/joca.2000.0369. PMID 11330253
- [Background] Blackburn J, Qureshi A, Amirfeyz R, Bannister G. Does preoperative anxiety and depression predict satisfaction after total knee replacement? Knee. 2012 Oct;19(5):522-4. doi: 10.1016/j.knee.2011.07.008. Epub 2011 Aug 16. PMID 21846588
- [Background] Brander V, Gondek S, Martin E, Stulberg SD. Pain and depression influence outcome 5 years after knee replacement surgery. Clin Orthop Relat Res. 2007 Nov;464:21-6. doi: 10.1097/BLO.0b013e318126c032. PMID 17603386
- [Background] Riddle DL, Wade JB, Jiranek WA, Kong X. Preoperative pain catastrophizing predicts pain outcome after knee arthroplasty. Clin Orthop Relat Res. 2010 Mar;468(3):798-806. doi: 10.1007/s11999-009-0963-y. Epub 2009 Jul 8. PMID 19585177
- [Background] Rolfson O, Dahlberg LE, Nilsson JA, Malchau H, Garellick G. Variables determining outcome in total hip replacement surgery. J Bone Joint Surg Br. 2009 Feb;91(2):157-61. doi: 10.1302/0301-620X.91B2.20765. PMID 19190046
- [Background] Stamenkovic DM, Rancic NK, Latas MB, Neskovic V, Rondovic GM, Wu JD, Cattano D. Preoperative anxiety and implications on postoperative recovery: what can we do to change our history. Minerva Anestesiol. 2018 Nov;84(11):1307-1317. doi: 10.23736/S0375-9393.18.12520-X. Epub 2018 Apr 5. PMID 29624026
- [Background] Xu J, Twiggs J, Parker D, Negus J. The Association Between Anxiety, Depression, and Locus of Control With Patient Outcomes Following Total Knee Arthroplasty. J Arthroplasty. 2020 Mar;35(3):720-724. doi: 10.1016/j.arth.2019.10.022. Epub 2019 Oct 18. PMID 31708293
- [Background] Yang MMH, Hartley RL, Leung AA, Ronksley PE, Jette N, Casha S, Riva-Cambrin J. Preoperative predictors of poor acute postoperative pain control: a systematic review and meta-analysis. BMJ Open. 2019 Apr 1;9(4):e025091. doi: 10.1136/bmjopen-2018-025091. PMID 30940757
- [Background] Kahlenberg CA, Nwachukwu BU, McLawhorn AS, Cross MB, Cornell CN, Padgett DE. Patient Satisfaction After Total Knee Replacement: A Systematic Review. HSS J. 2018 Jul;14(2):192-201. doi: 10.1007/s11420-018-9614-8. Epub 2018 Jun 5. PMID 29983663
- [Background] Acar HV. Acupuncture and related techniques during perioperative period: A literature review. Complement Ther Med. 2016 Dec;29:48-55. doi: 10.1016/j.ctim.2016.09.013. Epub 2016 Sep 13. PMID 27912957
- [Background] Alattas SA, Smith T, Bhatti M, Wilson-Nunn D, Donell S. Greater pre-operative anxiety, pain and poorer function predict a worse outcome of a total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2017 Nov;25(11):3403-3410. doi: 10.1007/s00167-016-4314-8. Epub 2016 Oct 12. PMID 27734110
- [Background] Eberhart L, Aust H, Schuster M, Sturm T, Gehling M, Euteneuer F, Rusch D. Preoperative anxiety in adults - a cross-sectional study on specific fears and risk factors. BMC Psychiatry. 2020 Mar 30;20(1):140. doi: 10.1186/s12888-020-02552-w. PMID 32228525
- [Background] Song B, Yang Y, Teng X, Li Y, Bai W, Zhu J. Use of pre-operative anxiety score to determine the precise dose of butorphanol for intra-operative sedation under regional anesthesia: A double-blinded randomized trial. Exp Ther Med. 2019 Nov;18(5):3885-3892. doi: 10.3892/etm.2019.8040. Epub 2019 Sep 23. PMID 31611935
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Kuzminskaite V, Kaklauskaite J, Petkeviciute J. Incidence and features of preoperative anxiety in patients undergoing elective non-cardiac surgery. Acta Med Litu. 2019;26(1):93-100. doi: 10.6001/actamedica.v26i1.3961. PMID 31281222
- [Background] Stuyt EB, Voyles CA. The National Acupuncture Detoxification Association protocol, auricular acupuncture to support patients with substance abuse and behavioral health disorders: current perspectives. Subst Abuse Rehabil. 2016 Dec 7;7:169-180. doi: 10.2147/SAR.S99161. eCollection 2016. PMID 27994492
- [Background] Furuse N, Shinbara H, Uehara A, Sugawara M, Yamazaki T, Hosaka M, Yamashita H. A Multicenter Prospective Survey of Adverse Events Associated with Acupuncture and Moxibustion in Japan. Med Acupunct. 2017 Jun 1;29(3):155-162. doi: 10.1089/acu.2017.1230. PMID 28736592
- [Background] Zhang J, Shang H, Gao X, Ernst E. Acupuncture-related adverse events: a systematic review of the Chinese literature. Bull World Health Organ. 2010 Dec 1;88(12):915-921C. doi: 10.2471/BLT.10.076737. Epub 2010 Aug 27. PMID 21124716
- [Background] Xu S, Wang L, Cooper E, Zhang M, Manheimer E, Berman B, Shen X, Lao L. Adverse events of acupuncture: a systematic review of case reports. Evid Based Complement Alternat Med. 2013;2013:581203. doi: 10.1155/2013/581203. Epub 2013 Mar 20. PMID 23573135
- [Result] Chen CC, Yang CC, Hu CC, Shih HN, Chang YH, Hsieh PH. Acupuncture for pain relief after total knee arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):31-6. doi: 10.1097/AAP.0000000000000138. PMID 25158837
- [Result] Karst M, Winterhalter M, Munte S, Francki B, Hondronikos A, Eckardt A, Hoy L, Buhck H, Bernateck M, Fink M. Auricular acupuncture for dental anxiety: a randomized controlled trial. Anesth Analg. 2007 Feb;104(2):295-300. doi: 10.1213/01.ane.0000242531.12722.fd. PMID 17242083
- [Derived] Kainkaryam P, Vincze S, Takata E, Secor E, Panza G, Walker A, Gallagher G, Bergner A, Finkel J, Kumar M, Witmer D, Shekhman M, Nagarkatti D. Open-Label Randomized Clinical Trial to Assess the Effects of Preoperative Acupuncture in High Anxiety Patients Undergoing Total Knee or Hip Arthroplasty. J Integr Complement Med. 2025 Feb;31(2):174-182. doi: 10.1089/jicm.2024.0314. Epub 2024 Oct 9. PMID 39383026

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on their high anxiety score (according to the validated Amsterdam Preoperative Anxiety and Information Scale (APAIS-A-T>10) who are scheduled for elective total knee or hip arthroplasty surgery at Bone and Joint Center from March 2022 to April 2023. The first patient was enrolled in March 21, 2022 and the last patient was enrolled in April 3, 2023.
Pre-assignment Details: Of 123 screened patients, 60 met the inclusion criteria and were randomized to treatment. 31 patients declined participation, 26 patients did not meet the eligibility criteria, 5 patients consented but had surgery cancellation, and 1 patient withdrew consent.
Groups:
- Acupuncture: Preoperative acupuncture
  Acupuncture needles: The acupuncture intervention includes a combination of auricular and body acupuncture. The auricular points used are Shen men, Zero point, Tranquilizer point, and Master cerebral.
  The body points used are the wrist PC6.
Period: Overall Study
Arm/Group | Acupuncture | Control
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Preoperative surveys missed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.60 (9.71) | 67.63 (7.71) | 68.62 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 47
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 26 | 29 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 26 | 24 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 32.16 (5.31) | 30.44 (5.51) | 31.30 (5.44)
Charlson Comorbidity Index (CCI) [Median (Inter-Quartile Range); unit: units on a scale] — Charlson Comorbidity Index is a morbidity score for mortality ris, it identifies 19 comorbidities and assigns weight to each, ranging from 1 to 6 points. The total score is the sum of points and ranges 0 (no disease burden) to 29 (maximal disease burden). Conditions are MI, CHF, PVD, cerebrovascular disease, dementia, chronic pulmonary disease, connective tissue disease, ulcer disease, mild liver disease, diabetes, hemiplegia, moderate or several renal disease, diabetes with end organ damage, any tumor, leukemia, lymphoma, moderate or severe liver disease, metastatic solid tumor, AIDS.
  units on a scale | 1.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
History of mental illness [Count of Participants; unit: Participants]
  History of mental illnesses | 15 | 12 | 27
  Anxiety | 13 | 10 | 23
  Bipolar disorder | 0 | 1 | 1
  Depression | 8 | 6 | 14
History of acupuncture [Count of Participants; unit: Participants]
  Yes | 12 | 7 | 19
  No | 18 | 23 | 41
Modified Amsterdam Pre-operative Anxiety and Information Scale (APAIS) Score [Mean (Standard Deviation); unit: units on a scale] — The Modified Amsterdam Pre-operative Anxiety and Information Scale (APAIS-A-T) is a modified survey that quantifies preoperative anxiety using four instead of six questions about anesthesia- and surgery-related anxiety, with each question scoring from 1 (not at all) to 5 (extremely). Total score is the sum of the four questions which ranges from 4 to 20, a minimum score of 11 was used as the most accurate cutoff to identify patients with high anxiety in this study.
  units on a scale | 13.27 (2.39) | 13.90 (2.56) | 13.58 (2.48)
Preoperative Visual Analogue Scale Score [Mean (Standard Deviation); unit: units on a scale] — The Preoperative Visual Analogue Scale VAS is a unidimensional measure of anxiety. It is a straight horizontal line of 100 mm in length, scores 0-100, with the right end (0) defined as the no anxiety and the left end (100) as the worst or extremely anxious. This scale was completed by patients and measured by researchers using a ruler.
  units on a scale | 60.73 (21.28) | 59.66 (30.11) | 60.20 (25.77)
Surgery type [Count of Participants; unit: Participants]
  Total Hip Arthroplasty | 15 | 16 | 31
  Total Knee Arthroplasty | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Perioperative Anxiety
Description: Determine the effect of preoperative acupuncture on preoperative anxiety in the acupuncture group using VAS (Visual Analog Scale) which is a 10 centimeters line in length, from 0-100, with 0 at the left extreme being "not at all anxious" and 100 at the right extreme being "very anxious". Participants put a cross on the line to indicate how they felt at the time point used. A higher score means worse as it means high anxiety.
Time Frame: Prior to acupuncture and 30 minutes after acupuncture
Population: Only participants in the acupuncture group (n=30) completed the Visual Analog Scale to reflect the level of anxiety they had before and 30 minutes after receiving the acupuncture procedure.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Preoperative Pre-acupuncture: Participants in the acupuncture group completed the Visual Analog Scale for anxiety immediately prior to having the acupuncture procedure
- Preoperative Post-acupuncture: Participants in the acupuncture group completed the Visual Analog Scale for anxiety 30 minutes after having the acupuncture procedure
Arm/Group | Preoperative Pre-acupuncture | Preoperative Post-acupuncture
Number analyzed (Participants) | 30 | 30
score on a scale | 60.73 (21.28) | 28.90 (21.54)
Statistical Analysis 1: Comparison: Preoperative Pre-acupuncture vs Preoperative Post-acupuncture; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Primary Outcome: Postoperative Pain in the First 3 Postoperative Hours
Description: Determine the effect of preoperative acupuncture on postoperative pain in both groups, using the self-reported NPS (Numeric Pain Scale) which is a scale of 0-10 where 0 is "no pain" and 10 is "severe pain". Using the mean pain score to compare the mean of the total pain in the first 3 postoperative hours between groups.
Time Frame: Total mean pain in the first 3 postoperative hours
Population: Total mean pain in the first 3 postoperative hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 1.93 (1.63) | 2.79 (2.83)
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.029, t-test, 2 sided

3. Secondary Outcome: Patient Satisfaction With Acupuncture Procedure
Description: Patients' satisfaction with acupuncture intervention was assessed in the acupuncture group only using the satisfaction scale of (1-5), where 1 is Extremely satisfied, 2 is Very satisfied, 3 is Somewhat satisfied, 4 is Not very satisfied, and 5 is Not at all satisfied. Each frequency represented the percentage of patients who were satisfied (given a score of 1 or 2 out of 5) with their acupuncture treatment. This assessment was done within a week after discharge, via a phone call.
Time Frame: Within 1 week after hospital discharge
Measure: Count of Participants; unit: Participants
Groups:
- Acupuncture Group: Patients who received the preoperative acupuncture procedure.
Arm/Group | Acupuncture Group
Number analyzed (Participants) | 30
Participants | 22

4. Secondary Outcome: Preoperative Pain
Description: Determine the effect of preoperative acupuncture on preoperative pain in the acupuncture group using the self-reported NPS (Numeric Pain Scale) which is a scale of 0-10 where 0 is "no pain" and 10 is "severe pain". Using the mean pain score to compare pre-acupuncture pain to post-acupuncture pain score in the acupuncture group only.
Time Frame: Prior to acupuncture and 30 minutes after acupuncture
Population: Only participants in the acupuncture group (n=30) completed the Numeric Pain Scale to reflect the level of pain they had before and 30 minutes after receiving the acupuncture procedure.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Preoperative Pre-acupuncture: Participants in the acupuncture group completed the Numeric Pain Scale immediately before having the acupuncture procedure
- Preoperative Post-acupuncture: Participants in the acupuncture group completed the Numeric Pain Scale 30 minutes after having the acupuncture procedure
Arm/Group | Preoperative Pre-acupuncture | Preoperative Post-acupuncture
Number analyzed (Participants) | 30 | 30
score on a scale | 4.97 (3.01) | 2.90 (6.62)
Statistical Analysis 1: Comparison: Preoperative Pre-acupuncture vs Preoperative Post-acupuncture; Test type: Superiority; p < 0.001, t-test, 2 sided

5. Secondary Outcome: Opioid Consumption
Description: Postoperative opioid consumption to be converted into morphine milliequivalents (MMEs) and compared between the two groups for up to 24 hours post surgery.
Time Frame: During hospitalization, up to 24 hours post surgery
Measure: Mean (Standard Deviation); unit: Morphine MilliEquivalent
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
Morphine MilliEquivalent | 45.51 (30.02) | 52.46 (30.92)
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.38, t-test, 2 sided

6. Secondary Outcome: Midazolam Use as Anxiolytic Medications
Description: The dose of Midazolam as an anxiolytic medication that was given at any time throughout hospitalization up to 24 postoperative hours.
Time Frame: During hospitalization, up to 24 hours post surgery
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
milligrams | 3.96 (1.73) | 4.21 (1.80)
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.61, t-test, 2 sided

7. Secondary Outcome: Patient Satisfaction Scale With Overall Care
Description: Patients' satisfaction with overall care management was compared using the patient satisfaction scale of (1-10), where 1 is extremely unsatisfied and 10 is extremely satisfied with overall care. Each frequency represents the percentage of patients in each group who have been either satisfied or extremely satisfied (given a score of 9 or 10 out of 10). This assessment was done within a week after discharge, via a phone call.
Time Frame: Within 1 week after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
Participants | 21 | 24
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.37, Chi-squared

8. Secondary Outcome: Occurrence of Nausea and Vomiting at First Postoperative Hour
Description: Compare the occurrence of postoperative nausea and vomiting using the Simplified Postoperative Nausea and Vomiting Impact Scale which consists of two questions, with a possible response total score of 0-6. Response score totals of 0-2 require no intervention. Response score totals of 3-4 may necessitate antiemetic medication. Response score totals of 5-6 are considered clinically important nausea requiring medication intervention, as this would constitute patients with excessive vomiting. This scale was used to report the occurrence of nausea (yes/no), with "yes" defined as any number above 0 in the scale, while "no" defined as 0.
Time Frame: At 1 postoperative hour
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
Participants
  Yes | 0 | 4
  No | 30 | 26
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.11, Fisher Exact

9. Secondary Outcome: Antiemetic Medications
Description: The frequency of any antiemetic medication given at any time throughout hospitalization up to 24 postoperative hours
Time Frame: During hospitalization, up to 24 hours post surgery
Measure: Median (Inter-Quartile Range); unit: number of doses
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
number of doses | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Hospital Length of Stay
Description: Using the hospital admission and discharge dates & times; this will be compared between the two groups.
Time Frame: From the date and time of admission to the date and time of discharge, assessed as 24-48 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
hours | 29.5 [27.8 to 31.3] | 29.0 [27.0 to 30.0]
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Postoperative Pain Upon Arrival to the PACU
Description: Determine the effect of preoperative acupuncture on postoperative pain in both groups, using the self-reported NPS (Numeric Pain Scale) which is a scale of 0-10 where 0 is "no pain" and 10 is "severe pain". Using the mean pain score to compare the mean pain scores between groups upon arrival to the PACU.
Time Frame: Postoperative pain at time of PACU arrival
Population: Mean pain scores upon arrival to the PACU between the groups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 0.47 (1.36) | 1.38 (2.83)
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.087, t-test, 2 sided

12. Secondary Outcome: Postoperative Pain at 1 Postoperative Hour
Description: Determine the effect of preoperative acupuncture on postoperative pain in both groups, using the self-reported NPS (Numeric Pain Scale) which is a scale of 0-10 where 0 is "no pain" and 10 is "severe pain". Using the mean pain score to compare the mean of pain scores at the first postoperative hour between groups.
Time Frame: At the first postoperative hour
Population: Using the mean of pain scores reported by participants at the first postoperative hour
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 1.67 (2.22) | 2.45 (3.15)
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.147, t-test, 2 sided

13. Secondary Outcome: Postoperative Pain After 3 Postoperative Hours
Description: Determine the effect of preoperative acupuncture on postoperative pain in both groups, using the self-reported NPS (Numeric Pain Scale) which is a scale of 0-10 where 0 is "no pain" and 10 is "severe pain". Using the mean pain score to compare the mean pain scores after three postoperative hours between groups.
Time Frame: After three postoperative hours
Population: Using the mean pain scores after three postoperative hours between groups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 3.67 (3.03) | 4.55 (3.29)
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.098, t-test, 2 sided

14. Secondary Outcome: Number of Participants That Received Midazolam Dose >2mg
Description: The number of participants who received a dose of midazolam exceeding 2 mg indicated a high level of perioperative anxiety that necessitated pharmacological intervention. The decision to use a dose higher than 2 mg was based on the standard practice of administering 2 mg of midazolam for preoperative regional nerve blocks; any dosage surpassing this amount was specifically intended for anxiety management.
Time Frame: During hospitalization up to 24 postoperative hours
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
Participants | 19 | 22
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.41, Chi-squared

15. Secondary Outcome: Patient's Satisfaction With Pain Management
Description: Patients' satisfaction with their postoperative pain management was compared between groups using the satisfaction scale of (1-10), where 1 is extremely unsatisfied and 10 is extremely satisfied. Each frequency represented the percentage of patients in each group who were satisfied (given a score of 9 or 10 out of 10)This assessment was done within a week after discharge, via a phone call.
Time Frame: Within 1 week after hospital discharge
Population: Each frequency represented the percentage of patients in the group who were satisfied (given a score of 9 or 10 out of 10)
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
Participants | 19 | 20
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.79, Chi-squared

16. Secondary Outcome: Patient's Satisfaction With Anxiety Management
Description: Patients' satisfaction with their perioperative anxiety management was compared between groups using the satisfaction scale of (1-10), where 1 is extremely unsatisfied and 10 is extremely satisfied. Each frequency represented the percentage of patients in each group who were satisfied (given a score of 9 or 10 out of 10). This assessment was done within a week after discharge, via a phone call.
Time Frame: Within 1 week after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
Participants | 21 | 19
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.58, Chi-squared

17. Secondary Outcome: Acupuncture Patients Who Were Likely to Consider Acupuncture for Future Surgeries
Description: Patients with acupuncture intervention were assessed for how likely to consider acupuncture for future surgeries using a scale of (1-4), where 1 is Very likely, 2 is Likely, 3 is Maybe, and 4 is Never. Each frequency represented the percentage of patients who were more likely (given a score of 1 or 2 out of 4) to receive acupuncture treatment in a future surgery. This assessment was done within a week after discharge, via a phone call.
Time Frame: Within 1 week after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture Group
Number analyzed (Participants) | 30
Participants | 25

18. Secondary Outcome: Occurrence of Nausea and Vomiting After 3 Postoperative Hours
Description: as for outcome 8
Time Frame: After 3 postoperative hours
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
Participants
  Yes | 5 | 5
  No | 25 | 25
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 1.00, Chi-squared

19. Secondary Outcome: Postoperative Pain in the First 3 Postoperative Hours (Group X Time)
Description: Determine the effect of preoperative acupuncture on postoperative pain in both groups, using the self-reported NPS (Numeric Pain Scale) which is a scale of 0-10 where 0 is "no pain" and 10 is "severe pain". To compare mean pain scores between groups, considering all 3 individual time points (at arrival to Post-Anesthesia Care Unit, 1st Postoperative hour, and 3rd Postoperative hour)
Time Frame: Mean pain scores at arrival to Post-Anesthesia Care Unit, 1st Postoperative hour, and 3rd Postoperative hour
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 30 | 30
score on a scale
  at arrival to PACU | 0.47 (1.36) | 1.38 (2.83)
  1hr post-operation | 1.67 (2.22) | 2.45 (3.15)
  3hr post-operation | 3.67 (3.03) | 4.55 (3.29)
Statistical Analysis 1: Comparison: Acupuncture vs Control; Test type: Superiority; p = 0.919, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 30 postoperative days
Groups:
- Control Group: Patients who did not receive the preoperative acupuncture procedure.
Arm/Group | Acupuncture Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 13/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acupuncture Group (N=30) | Control Group (N=30)
Local bleeding (Surgical and medical procedures) | 9 (9) | 0 (0) — Immediate complication of acupuncture which is a few drops of blood at the site of the acupuncture needle insertion
Discomfort (Surgical and medical procedures) | 1 (1) | 0 (0) — Discomfort during the acupuncture procedure
Residual pain (Surgical and medical procedures) | 3 (3) | 0 (0) — Mild pain after removing the acupuncture needles

LIMITATIONS AND CAVEATS:
The limitation of this study is the open-label aspect could be associated with placebo effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT06099223/Prot_SAP_ICF_000.pdf